CLINICAL TRIAL: NCT04099992
Title: Sympatho-inhibition With Mindfulness in Chronic Kidney Disease (MIND-CKD)
Brief Title: Mindfulness in Chronic Kidney Disease
Acronym: MIND-CKD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jeanie Park, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00110956; 5R61AT010457 (NIH); 4R33AT010457 (NIH)
Record Dates: First submitted 2019-09-20; First posted 2019-09-23 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Chronic Kidney Diseases
Keywords: Mindfulness; Transcutaneous Vagus Nerve Stimulation; tVNS; Sympatho-inhibitory effects
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Protocol 1 (R61): 50 CKD participants will be randomized to MBSR (N=25) versus an active control intervention (health enhancement program; N=25).
  Protocol 2 (R33): 100 CKD participants will be randomized to MBSR+tVNS (n=25), MBSR+sham-tVNS (n=25), HEP+tVNS (n=25), and HEP+sham-tVNS (n=25).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A third-party investigator outside of the research team will label both real and sham devices with a coded number so that both participants and investigators can remain double-masked during the clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Mindfulness-Based Stress Reduction (MBSR) (Experimental): Mindfulness-Based Stress Reduction (MBSR) tis designed to provide education about mindfulness and stress; experiential mindfulness practice, and discussion of participants' experiences with mindfulness practice. MBSR is delivered in 8 weekly 2.5-hour group sessions and one day-long retreat that occurs after the 6th session.
  Interventions: Behavioral: Mindfulness-based stress reduction (MBSR)
- Health enhancement program (HEP) (Active Comparator): Health enhancement program (HEP) is designed to provide a structurally parallel, active control intervention to MBSR with health benefits in their own right, while omitting any components of mindfulness. HEP participants will meet with a health educator in a group setting for 8 weekly 2.5-hour sessions with a day-long retreat.
  Interventions: Behavioral: Health enhancement program (HEP)
- MBSR+tVNS (Experimental): Mindfulness-Based Stress Reduction (MBSR) tis designed to provide education about mindfulness and stress; experiential mindfulness practice, and discussion of participants' experiences with mindfulness practice. MBSR is delivered in 8 weekly 2.5-hour group sessions and one day-long retreat that occurs after the 6th session.
  Transcutaneous vagus nerve stimulation (tVNS) is a simple, noninvasive, self-administered adjunctive therapy, that may enhance the sympatho-inhibitory effects of mindfulness meditation (MM) in chronic kidney disease (CKD) .
  Interventions: Behavioral: Mindfulness-based stress reduction (MBSR); Device: Transcutaneous Vagus Nerve Stimulation (tVNS)
- MBSR+sham-tVNS (Active Comparator): Mindfulness-Based Stress Reduction (MBSR) tis designed to provide education about mindfulness and stress; experiential mindfulness practice, and discussion of participants' experiences with mindfulness practice. MBSR is delivered in 8 weekly 2.5-hour group sessions and one day-long retreat that occurs after the 6th session.
  Sham stimulation will be delivered using a sham device that is identical in appearance and function to tVNS, but programmed to produce a lower frequency biphasic signal that can be felt by the participant without actually stimulating the vagus nerve.
  Interventions: Behavioral: Mindfulness-based stress reduction (MBSR); Device: Sham-transcutaneous Vagus Nerve Stimulation (tVNS)
- HEP+tVNS (Experimental): Health enhancement program (HEP) is designed to provide a structurally parallel, active control intervention to MBSR with health benefits in their own right, while omitting any components of mindfulness. HEP participants will meet with a health educator (a registered dietician) in a group setting for 8 weekly 2.5-hour sessions.
  Transcutaneous vagus nerve stimulation (tVNS) is a simple, noninvasive, self-administered adjunctive therapy, that may enhance the sympatho-inhibitory effects of mindfulness meditation (MM) in chronic kidney disease (CKD).
  Interventions: Behavioral: Health enhancement program (HEP); Device: Transcutaneous Vagus Nerve Stimulation (tVNS)
- HEP+sham-tVNS (Active Comparator): Health enhancement program (HEP) is designed to provide a structurally parallel, active control intervention to MBSR with health benefits in their own right, while omitting any components of mindfulness. HEP participants will meet with a health educator in a group setting for 8 weekly 2.5-hour sessions.
  Sham stimulation is be delivered using a sham device that is identical in appearance and function to tVNS, but programmed to produce a lower frequency (0.1 Hz) biphasic signal that can be felt by the participant without actually stimulating the vagus nerve.
  Interventions: Behavioral: Health enhancement program (HEP); Device: Sham-transcutaneous Vagus Nerve Stimulation (tVNS)

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction (MBSR) — Mindfulness-based stress reduction (MBSR) is delivered in 8 weekly 2.5-hour group sessions and one day-long retreat that occurs after the 6th session. MBSR teaches to become more aware of thoughts, feelings, and sensations, and to skillfully respond to stressors. Each of the sessions includes education about mindfulness and stress; experiential mindfulness practice, and discussion of participants' experiences with mindfulness practice. Participants learn formal mindfulness practices (e.g., meditation, yoga, body scan, body scan) as well as informal such as awareness of breath, thoughts, or emotions, and mindfulness of daily activities. Participants will receive digital audio (MP3) downloads with guided MM practices, a home practice manual, and handouts with each week's assignments. Daily home practice will consist of 40-45 minutes of recorded practice. Participants will log their daily practice. If a participant misses a class, it is possible to make up the class on a different day.
  Arms: MBSR+sham-tVNS; MBSR+tVNS; Mindfulness-Based Stress Reduction (MBSR)
Behavioral: Health enhancement program (HEP) — 8-week health enhancement program (HEP) is designed to provide a structurally parallel, active control intervention to MBSR with health benefits in their own right, while omitting any components of mindfulness. HEP matches MBSR in structure and content, and in parallel to MBSR, consists of music therapy, nutritional education, posture and balance movements, walking and stretching. Work with all practices with group discussion and exercises during an all-day "spa day" will match the all-day retreat in MBSR. HEP participants will meet with a health educator in a group setting for 8 weekly 2.5-hour sessions. Participants will receive MP3 downloads on an MP3 player with recordings of health education topics, a home listening manual, and weekly handouts with each week's listening assignments. Participants will listen to these MP3 recordings daily for 40-45 minutes and log their daily adherence.
  Arms: HEP+sham-tVNS; HEP+tVNS; Health enhancement program (HEP)
Device: Transcutaneous Vagus Nerve Stimulation (tVNS) — Participants self-administer tVNS twice per day for 8 weeks. tVNS is delivered using a multi-use, hand-held, rechargeable portable device consisting of a rechargeable battery, signal generating and amplifying electronics, and a button for operator control of the stimulation intensity. Conductive gel is applied to the stainless steel round discs on the device and placed vertically on the skin overlying the vagus nerve under the angle of the mandible, between the trachea and sternocleidomastoid muscle. A low-voltage electrical signal is delivered consisting of 5-kilohertz (kHz) sine wave series for 1 ms and repeated every 40 ms, with a maximum delivery of 24 V and 60 milliampere (mA) output. Stimulation amplitude is adjusted by the user and is increased until there is a vibration and slight muscle contraction in the lower face or neck. Stimulation is delivered for 2 minutes on the left side of the neck, and 2 minutes on the right side of the neck, for a total 4 minutes per one dose.
  Other Names: gammaCore; Electrocore
  Arms: HEP+tVNS; MBSR+tVNS
Device: Sham-transcutaneous Vagus Nerve Stimulation (tVNS) — Participants self-administer sham-tVNS twice per day for 8 weeks. Sham stimulation will be delivered using a sham device that is identical in appearance and function, but programmed to produce a lower frequency biphasic signal that can be felt by the participant without actually stimulating the vagus nerve.
  Arms: HEP+sham-tVNS; MBSR+sham-tVNS

SUMMARY:
This study will test whether mindfulness meditation (MM) improves sympathetic function in chronic kidney disease (CKD) and whether transcutaneous vagus nerve stimulation (tVNS) optimizes the sympatho-inhibitory effects of mindfulness meditation (MM) and restores autonomic balance in CKD patients.

DETAILED DESCRIPTION:
Approximately 30 million people in the US have chronic kidney disease (CKD) and are at 5-15 fold greater risk of cardiovascular (CV) disease and mortality. A major factor contributing to increased CV risk in these patients is chronic elevation of sympathetic nervous system (SNS) activity.

Patients with even minimal decrements in kidney function have significant and substantial increases in SNS activity and reactivity that are independently linked to adverse CV events. The mechanisms underlying SNS overactivity in CKD are multifactorial, and include chronic inflammation and blunted arterial baroreflex sensitivity (BRS). SNS overactivity, in turn, leads to downstream deleterious effects on ambulatory BP profiles characterized by higher daytime BP, and lack of normal reductions in nocturnal BP (i.e. nocturnal nondipping), both of which are independently linked to increased CV risk. Current treatments to combat SNS overactivity are limited to sympatholytic medications such as β-blockers, α-blockers, and clonidine; however, these pharmacologic agents are associated with long-term adverse metabolic consequences such as insulin resistance and hyperlipidemia, and often intolerable side effects such as fatigue, orthostatic hypotension, and rebound hypertension. New therapeutic strategies to safely and effectively ameliorate SNS over-activity are of paramount importance to improve clinical outcomes in this highly prevalent and high-risk patient population.

Mindfulness meditation (MM) may be one such novel, safe, and effective approach at improving hemodynamics and autonomic function in CKD. Prior studies have shown that 8 weeks of mindfulness-based stress reduction (MBSR) lowers BP in a variety of patient groups. Although the mechanisms are poorly understood, studies using indirect measures of SNS activity such as heart rate variability suggest that MM may exert its hemodynamic effects via autonomic modulation.

This study tests whether mindfulness meditation (MM) improves sympathetic function in chronic kidney disease (CKD) and whether transcutaneous vagus nerve stimulation (tVNS) optimizes the sympatho-inhibitory effects of mindfulness meditation (MM) and restores autonomic balance in CKD patients. These study aims are tested with two separate protocols.

Protocol 1 tests the sustained effects of MBSR on SNS function and BP profiles in CKD. Participants will be randomized to 8 weeks of MBSR or a health enhancement program (HEP).

Protocol 2 tests an optimization strategy to enhance the sympatho-inhibitory effects of MM and restore autonomic balance using transcutaneous vagus nerve stimulation (tVNS) in CKD. The vagus nerve, the major effector of the parasympathetic nervous system (PNS), is composed of afferent nerve fibers that connect to the nucleus tractus solitarii (NTS) and other brainstem regions that influence central SNS output and baroreflexes, and efferent nerve fibers that activate the cholinergic anti-inflammatory pathway. Both experimental and human studies have shown promising results that stimulation of the vagus nerve lowers BP reduces SNS activity, improves BRS, and lowers inflammation. Participants with Stage III and IV CKD will be randomized into one of four study arms: MBSR with tVNS, MBSR with sham-tVNS, HEP with tVNS, and HEP with sham-tVNS. Participants will self-administer tVNS or sham-tVNS twice per day for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* stages III and IV CKD as defined by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation
* stable renal function (no greater than a decline of eGFR of 1 cc/min/1.73 m2 per month over the prior 3 months)

Exclusion Criteria:

* severe CKD (eGFR<15 cc/min)
* diabetic neuropathy
* autonomic dysfunction
* any serious disease that might influence survival
* anemia with hemoglobin <10 g/dL
* treatment with central α-agonists or monoamine oxidase (MAO) inhibitors
* myocardial infarction or cerebrovascular accident within the past 6 months
* uncontrolled hypertension (BP≥170/100 mm Hg)
* low BP (BP<100/50 mm Hg)
* bradycardia (HR<55 beats/min)
* ongoing drug or alcohol abuse (defined as >2 drinks/day in men, and >1 drink/day in women)
* surgery within the past 3 months
* adjustment of antihypertensive medications within the past month
* pregnancy or plans to become pregnant
* psychosis
* suicidal ideation
* implanted electronic or metallic device such as a pacemaker
* implanted hearing aid, bone plate, carotid stent, bone screw at or near the neck
* carotid atherosclerosis
* concurrent use of another stimulating device such as a transcutaneous electrical nerve stimulation (TENS) unit

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Mean Muscle Sympathetic Nerve Activity (MSNA) Burst Frequency (BF) | Baseline, 8 weeks
  Multiunit postganglionic sympathetic nerve activity is recorded from a tungsten microelectrode inserted into the peroneal nerve with a reference microelectrode inserted in close proximity. Efferent nerve signals are amplified, filtered, rectified and integrated (time constant 0.1 s) to obtain a mean voltage display of MSNA. MSNA bursts are automatically detected using the following criteria: burst-to-noise ratio of 3:1 within a 0.5-s search window, with an average latency of 1.2-1.3 s in burst occurrence from the previous R-wave. MSNA is expressed as burst frequency measured a bursts per minute.

SECONDARY OUTCOMES:
Change in Daytime Blood Pressure (BP) | Baseline, 8 weeks
  Blood pressure is assessed with 24-hour ambulatory BP monitoring. Upper arm readings will be taken for at least 24 hours. BP measurements will be made every 20 minutes during the daytime period, from 7 ante meridiem (AM) to 11 post meridiem (PM). Participants will record their wake and sleep times, and analyses will be adjusted for the participant's individual wake and sleep times.
Change in Nocturnal Dipping of Blood Pressure (BP) | Baseline, 8 weeks
  Blood pressure is assessed with 24-hour ambulatory BP monitoring. Upper arm readings will be taken for at least 24 hours. BP measurements will be made every 30 minutes during the nighttime period, from 11 PM to 7 AM. Participants will record their wake and sleep times, and analyses will be adjusted for the participant's individual wake and sleep times.
Change in Heart Rate Assessed by 24-hour EKG Monitoring | Baseline, 8 weeks
  The 24-hour EKG monitoring will be performed using a portable Holter monitor. Stickers will be placed on the participants chest to record their heart rate.
Change in Baroreflex Sensitivity (BRS) Among Protocol 2 Participants | Baseline, 8 weeks
  Afferent sympathetic baroreflex input travels to the brainstem via the glossopharyngeal and vagus nerves and integrate with brainstem centers that regulate efferent SNS (sympathetic BRS) and parasympathetic (cardiovagal BRS) outflow. BRS is defined as the change in interbeat interval (IBI) in milliseconds per unit change in BP. For example, when the BP rises by 10 mmHg and IBI increases by 100 ms, BRS would be 100/10 = 10 ms/mmHg.
Change in Tumor Necrosis Factor (TNF) Level Among Protocol 2 Participants | Baseline, 8 weeks
  Tumor necrosis factor (TNF) is a cell signaling protein (cytokine) involved in systemic inflammation and is one of the cytokines that make up the acute phase reaction. It will be measured by blood test.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanie Park, Principal Investigator — Emory University
Locations (1):
- Atlanta VA Medical Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article after deidentification (text, tables, figures, and appendices) will be available for sharing.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available for sharing beginning 9 months and ending 36 months following article publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal for individual participant data meta-analyses and whose proposed use of the data has been approved by an independent review committee identified for this purpose. Requests should be directed to Jeanie.park@emory.edu.